CLINICAL TRIAL: NCT00975208
Title: Osteogenesis and Dental Eruption Through Electrical Stimuli Following Periosteoplasty for Alveolar Clefts in Patients With Cleft Lip and Palate Deformities. A Preliminary Report.
Brief Title: Osteogenesis and Dental Eruption Through Electrical Stimuli
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of Guadalajara (Other)
Responsible Party: Christian Weigand, M.D., Instituto Jalisciense de Cirugía Reconstructiva de Jalsico, México
Other Study IDs: CW1234
Record Dates: First submitted 2009-09-10; First posted 2009-09-11 (Estimated); Last update posted 2009-09-11 (Estimated); Status verified 2009-09

CONDITIONS: Cleft Lip
Keywords: Osteogenesis [G07.700.320.500.325.377.625.100.729]; Tooth Eruption [G10.549.235.726]
MeSH Terms: conditions — Cleft Lip

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The closure of the alveolar cleft as part of cleft lip and palate deformities is a procedure that, to this date, still demands great efforts from plastic surgeons. The feasibility of periosteoplasty for reconstruction of the alveolar arcade as well as the use of electrical stimulation in order to increase osteoneogenesis have been proven in the past. The present study attempts to combine both procedures that have only been reported separately worldwide. The objective of this study is to increase the osteogenic capacity and hence, dental eruption.

ELIGIBILITY:
Inclusion Criteria:

* Patients with unilateral cleft lip and palate deformities and alveolar defects

Exclusion Criteria:

* Patients without alveolar cleft
* Patients with syndromes that did not require periosteoplastic procedures as well as patients with systemic illnesses that may affect the result of the study (for instance diabetes)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients of the Institute of Reconstructive Surgery of Jalisco, México
Sampling Method: Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2006-01; Primary Completion 2007-11 (Estimated); Study Completion 2010-08 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: José Guerrerosantos, M.D., Ph.D., Study Chair — Instituto Jalisciense de Cirugía Reconstructiva "Dr. Guerrerosantos"